CLINICAL TRIAL: NCT06732973
Title: A Randomized, Open- Label, Parallel Controlled Study to Compare the Pharmacokinetics of JS005 With a Pre-filled Syringe and a Pre-filled Automatic Syringe Subcutaneously Injected in Healthy Volunteers
Brief Title: A Bioequivalence Study of JS005 Pre-filled Syringe and JS005 Auto-injector
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS005-007-BE
Record Dates: First submitted 2024-12-02; First posted 2024-12-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Health Volunteer

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental：JS005 AI (Experimental): The drug was administered by a single subcutaneous injection via AI
  Interventions: Drug: JS005
- Experimental：JS005 PFS (Active Comparator): The drug was administered by a single subcutaneous injection via PFS
  Interventions: Drug: JS005

INTERVENTIONS:
Drug: JS005 — JS005：The drug was administered by a single subcutaneous injection

SUMMARY:
This study is a single-center, randomized, open-label, single-dose, parallel-controlled trial design conducted in healthy adult subjects. After signing the informed consent form and completing the screening examination, if the subjects meet all the inclusion criteria and do not meet any exclusion criteria, they will be randomly assigned to treatment group A or treatment group B: treatment group A receives a single subcutaneous injection of JS005 300 mg through PFS, and treatment group B receives a single subcutaneous injection of JS005 300 mg through AI. Subjects were followed up until the 85th day of the study to evaluate the pharmacokinetic equivalence of JS005. 136 subjects are planned to be included in each group.

The entire study cycle includes a screening period of up to 21 days and a follow-up period of 12 weeks (85 days). Subjects will be admitted to the Phase I clinical research ward on the day before administration (D-1), and can only leave after completing all examinations and evaluations on the 11th day after administration. They will return to the clinical research center for follow-up on days 15, 22, 29, 43, 57, 71, and 85.

ELIGIBILITY:
Inclusion criteria:

* Subjects voluntarily sign informed consent before any study-related procedures begin, are able to communicate smoothly with the investigator, understand and are willing to strictly comply with the clinical research protocol, study procedures, visit plans, treatment plans, laboratory tests, and other research requirements specified in the protocol.
* Healthy male or female volunteers aged 18 to 49 (inclusive);
* Body mass index (BMI) within the range of 18 to 26 kg/m2 (inclusive), with male weight ≥ 50kg and female weight ≥45kg.
* Female subjects with fertility, as well as significant other male subjects of childbearing age, must be willing to use high-efficiency contraceptive methods during the study period until 20 weeks (expected 5 half-lives) after the last study drug administration (see Annex 3). Female subjects with fertility must have negative pregnancy tests during the screening period and before randomization.

Exclusion Criteria:

* Previously used Secukinumab, Ixekizumab, Brodalumab, and other targeted drugs that directly act on IL-17 or IL-17 receptors.
* Any medication used within 2 weeks before randomization or the medication used on the day of randomization is still in the elimination period (within 5 half-lives), based on the length of time (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, etc.; excluding topical medication, female contraceptives, and regular vitamins);
* Those who have participated in any clinical trial of a drug or medical apparatus within 3 months before randomization, or those who are still in the follow-up period of a clinical study or within 5 half-lives of the trial drug (whichever is longer) before randomization. Participants in clinical trials are defined as those who have given informed consent to the clinical trial and have used the trial drug (including placebo) or the trial medical apparatus.
* Have a history of allergies to any research drug ingredients. Known allergies or hypersensitivity reactions to any biological therapy during screening, if participating in this study, will pose unacceptable risks to the subjects.
* Individuals with clear diseases of the Central Nervous System, cardiovascular system, digestive system, respiratory system, urinary system, hematological system, endocrine and metabolic systems, etc. that require medical intervention or other diseases that are not suitable for clinical trials (such as a history of mental illness, etc.) (within 5 years before screening).
* Those who have a history of blood donation in the past month, or have suffered severe blood loss (total blood volume ≥ 400 mL), or have received blood transfusions in the past 2 months.
* Within the first three months of randomization, smokers and alcoholics (drinking 14 units of alcohol per week: 1 unit = 360 mL of beer, or 45 mL of Baijiu, or 150 mL of wine; smoking > 5 cigarettes per day).
* History of Drug Abuse, or positive urine drug screening test during the screening period;
* Hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (Anti-HCV), Treponema pallidum antibody and acquired immunodeficiency syndrome (HIV) antibody positive;
* The medical history, symptoms, and examination results of the subjects suggest active or latent tuberculosis. The tuberculosis status of all subjects will be screened through gamma interferon release test (IGRA) and chest X-ray.Those who test positive for IGRA will be excluded.If the IGRA result is uncertain, re-testing is allowed. Subjects with uncertain results from both tests will be excluded from the study.Subjects who underwent IGRA and X-ray examinations within one month before randomization may not undergo IGRA and X-ray examinations again during the screening period, according to the researcher's judgment.
* Randomized individuals who have had severe trauma or undergone major surgery within the previous 6 months, or plan to undergo surgery during the trial period.
* Screening or base line vital signs, physical examination, clinical laboratory examination [blood routine, blood biochemistry, urine routine, coagulation function, gamma interferon release test (IGRA), blood pregnancy], electrocardiogram examination, abdominal B-ultrasound, chest X-ray examination with abnormalities and clinical.
* Random pre-glomerular filtration rate (eGFR) < 90 mL/min/1.73m2
* Random pre-alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or gamma-glutamyltransferase (GGT) exceeding 2 times ULN, or total bilirubin exceeding 1.5 times ULN
* Those with abnormal and clinically significant results in the first 12-lead electrocardiogram (e.g. male QTcF > 450ms, female QTcF > 470 ms; QTcF correction calculation using Fridericia formula, Fridericia formula: QTcF = QT/(RR ^ 0.33), RR is the standardized heart rate value, obtained by dividing 60 by heart rate).
* Pregnant or lactating women or male subjects whose spouses have pregnancy plans during the study period.
* Subjects who have been vaccinated or exposed to any live or attenuated vaccine within the previous 6 weeks of randomization, or who are expected to receive the above vaccines during study treatment or within 8 weeks after study drug discontinuation.
* Researchers believe that there are other factors that are not suitable for participating in the experiment.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 272 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
AUC0-last | 85 days
  Area under the time-concentration curve from time 0 to last time of quantifiable concentration
Cmax | 85 days
  Maximum Concentration
AUC0-inf | 85 days
  Area under the time-concentration curve from time 0 to inf of quantifiable concentration

SECONDARY OUTCOMES:
incidence and severity of adverse events(AE) | 85 days
  incidence and severity of adverse events(AE)
The time to reach Cmax （Tmax） | 85 days
  Pharmacokinetic (PK) parameters of JS005 :The time to receive reach Cmax （Tmax）
Apparent clearance(CL/F) | 85 days
  Apparent clearance(CL/F) of JS005 :apparent clearance(CL/F)
T1/2 | 85 days
  Elimination half-life of JS005
Vz/F | 85 days
  Apparent volume of distribution of JS005
ADA | 85 days
  Incidence of anti-JS005 drug antibodies (ADA)
ADA-positive | 85 days
  Titers of ADA-positive samples
NAb | 85 days
  Incidence of neutralizing antibodies (NAb)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengzhou Sixth People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided